CLINICAL TRIAL: NCT03705247
Title: The Role of Bleeding at Implant Placement: a Prospective Observational Study
Brief Title: The Role of Bleeding at Implant Placement
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S58575
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2018-10

CONDITIONS: Bleeding; Angiogenesis; Peri-Implantitis
Keywords: Dental Implants
MeSH Terms: conditions — Hemorrhage; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Angiogenesis is inherently associated to bone formation and healing. During implant osseointegration, a successive and successful angiogenic processes has to occur to promote bone formation. In 1969, Branemark et al. demonstrated that direct contact between bone and titanium implant surface was possible, defining osseointegration as "the direct, structural, and functional contact between live bone and the surface of a functionally loaded implant". Consequently, the need of an empirical measurement appeared. With the introduction of resonance frequency analysis (RFA), it is now possible to measure the degree of implant stability at any time during the course of implant treatment and loading. In this way, changes in implant stability can be monitored over the time and it is likely possible to find implants at risk of failure before they become loose. The rationale of this study is to analyse how important a good vascularization is for the future bone formation around dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Males or females American Society of Anesthesiologists classification (ASA) I or II, between 18 to 80 years of age
* Patient in good general health as documented by self-assessment.
* Patients needing implant rehabilitation in the upper or lower jaw.
* Patients must be committed to the study and must be willing to sign the informed consent.

Exclusion Criteria:

* Any systemic medical condition that could interfere with the surgical procedure or planned treatment.
* Immunosuppression, Diabetes, Anticoagulation or Antiaggregatory medication.
* Current pregnancy or breast feeding/ lactating at the time of recruitment.
* Radiotherapy or Chemotherapy in head and neck area.
* Intravenous and oral bisphosphonate therapy.
* Patients smoking >20 cigarettes a day.
* Unwillingness to return for the follow-up examination.
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unrealistic expectations.

Local exclusion criteria:

* Immediate implant placement after tooth extraction.
* Risk of extra bleeding due to inflammatory or infectious processes near the zone of implantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who come to the Unit of Periodontology (UZ Leuven, St. Rafaël), in need of implant rehabilitation, will be evaluated for initial study eligibility during a screening visit. Patients shall be advised of the need to attend follow-up visits: 3 months after implant placement (at abutment placement visit) and 1 year, the latter to analyse the early bone remodelling.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Correlation between bleeding during implant placement and marginal bone loss | 1 year
  Peri-implant bone loss after 1 year from the implant placement

SECONDARY OUTCOMES:
Correlation between bleeding during implant placement and implant stability quotient (ISQ) values | 3 months
  Correlation between bleeding during implant placement and implant stability quotient (ISQ) values

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium